CLINICAL TRIAL: NCT00787787
Title: The CapSul Trial: A Phase II Study of Sunitinib and Capecitabine for the Treatment of Unresectable or Metastatic Hepatocellular Carcinoma (HCC)
Brief Title: Sunitinib Malate and Capecitabine in Treating Patients With Unresectable or Metastatic Liver Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6553; NCI-2010-00605 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-04

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sunitinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (sunitinib malate and capecitabine) (Experimental): Patients receive sunitinib malate PO QD on days 1-21 and capecitabine PO BID on days 1-14. Courses repeat every 21 days in the absence or disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate; Drug: capecitabine

INTERVENTIONS:
Drug: sunitinib malate — Given PO
  Other Names: SU11248; sunitinib; Sutent
Drug: capecitabine — Given PO
  Other Names: CAPE; Ro 09-1978/000; Xeloda

SUMMARY:
This phase II trial studies how well giving sunitinib malate together with capecitabine works in treating patients with unresectable or metastatic liver cancer. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sunitinib malate together with capecitabine may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression-free survival of patients with unresectable or metastatic hepatocellular carcinoma (HCC) treated with sunitinib and capecitabine.

SECONDARY OBJECTIVES:

I. To determine the overall survival, response rate by Response Evaluation Criteria in Solid Tumors (RESIST) criteria, alpha fetoprotein (AFP) response, survival at one year, and safety and tolerability.

OUTLINE:

Patients receive sunitinib malate orally (PO) once daily (QD) on days 1-21 and capecitabine PO twice daily (BID) on days 1-14. Courses repeat every 21 days in the absence or disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of hepatocellular carcinoma (HCC) OR meets radiographic criteria for diagnosis of HCC without biopsy
* Liver mass at least 1 cm up to 2 cm in size: classic enhancement on 2 approved imaging modalities
* Liver mass > 2 cm in size: classic enhancement on 1 approved imaging modality
* At least one site of bidimensional measurable disease with the longest axis >= 20mm by conventional computed tomography (CT) scan or >= 10mm by spiral CT scan or >= 10mm by magnetic resonance imaging (MRI)
* Not eligible for curative intent surgery and not eligible for, or not willing to undergo, orthotopic liver transplantation
* Patient has received =< 1 prior systemic therapy
* Patient has completed treatment with surgery at least 4 weeks prior to study drug administration
* Patient has completed other cancer directed treatments including systemic chemotherapy, transarterial chemotherapy, transarterial chemoembolization or bland embolization, targeted therapy, radiotherapy, or treatment with other investigational anti-cancer agents at least 4 weeks prior to study drug administration AND has radiographic evidence of disease progression following these treatments
* Life expectancy of greater than 12 weeks
* Child-Pugh class A or B
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Karnofsky > 60%)
* Platelet count >= 75,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) =< 5 times upper limit of normal (ULN)
* Total bilirubin =< 3 times ULN
* Calculated or measured creatinine clearance >= 40 mL/min
* Prothrombin time =< 1.5 international normalized ratio (INR)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document and comply with scheduled visits, treatment plan, laboratory testing, and other trial procedures

Exclusion Criteria:

* History of another cancer within the last 5 years with the exception of localized basal or squamous cell carcinoma of the skin or stage 1A cervical cancer
* Known brain metastases, spinal cord compression, or evidence of symptomatic brain or leptomeningeal carcinomatosis on screening CT or MRI scan
* National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 Grade 2 variceal bleed within 6 weeks of registration or Grade 3 other bleed within 4 weeks of registration
* Any of the following within the 6 months prior to registration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
* Ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 Grade 2
* Prolonged QTc interval on baseline electrocardiograph (EKG)
* Uncontrolled Hypertension (> 150/100 mm Hg despite optimal medical therapy)
* Severe hepatic impairment, defined as Childs-Pugh Class C
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* Concurrent treatment on another clinical trial; supportive care trials or non-treatment trials, e.g. quality of life (QOL), are allowed
* Pregnancy or breastfeeding; female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy; all female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment; male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy; the definition of effective contraception will be based on the judgment of the principal investigator or a designated associate
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib or capecitabine

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-09; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Whiting, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to the lack of apparent benefit, the study was closed to further enrollment after the 7th patient was enrolled.
Period: Overall Study
Arm/Group | Treatment (Sunitinib Malate and Capecitabine)
Started | 7
Completed | 0
Not Completed | 7
Not completed — Lack of Efficacy | 4
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Sunitinib Malate and Capecitabine)
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 57 [28 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival
Description: Analyzed using the Kaplan-Meier method. Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). Progressive disease (PD) indicates at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From the start of treatment to time of progression or death from any cause, assessed up to 3 years
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Sunitinib Malate and Capecitabine)
Number analyzed (Participants) | 7
days | 203 [13 to 292]

2. Secondary Outcome: Best Response by RECIST Criteria
Description: Incidence rate of best clinical response (complete response [CR], partial response [PR], stable disease [SD], or progressive disease[PD]) as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST v1.0). CR indicates disappearance of all target lesions. PR indicates at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive disease indicates at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) indicates neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: From the start of the treatment until disease progression/recurrence, assessed every 3 months, up to 3 years
Population: Only 4 patients in this study had assessments of response by RECIST criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sunitinib Malate and Capecitabine)
Number analyzed (Participants) | 4
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 4

3. Secondary Outcome: Median Overall Survival
Description: Survival estimated by Kaplan-Meier method
Time Frame: From start of treatment until death from any cause, assessed up to 3 years
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Sunitinib Malate and Capecitabine)
Number analyzed (Participants) | 7
days | 282 [157 to 400]

ADVERSE EVENTS:
Time Frame: Day of first administration of study drugs to 30 days after last dose of study drug, up to 3 years.
Arm/Group | Treatment (Sunitinib Malate and Capecitabine)
All-Cause Mortality (participants affected / at risk) | 7/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sunitinib Malate and Capecitabine) (N=7)
Extrapyramidal myelinosis (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sunitinib Malate and Capecitabine) (N=7)
Headache (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hand-foot Syndrome (Skin and subcutaneous tissue disorders) | 5 (11)
Mucositis (Gastrointestinal disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (6)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Neutropenia (Blood and lymphatic system disorders) | 3 (10)
Hypertension (Vascular disorders) | 1 (1)
Oral Herpes Simplex infection (Infections and infestations) | 1 (1)
Thickened callus on foot (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Increased alanine amino transferase (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes